CLINICAL TRIAL: NCT01706185
Title: Analysis of the Incidence of Expression of Tumor Antigens in Cancer Tissue From Patients With Pathologically Demonstrated Bladder Cancer
Brief Title: Incidence of Expression of Tumor Antigens in Cancer Tissue From Patients With Pathologically Demonstrated Bladder Cancer
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111294
Record Dates: First submitted 2012-10-04; First posted 2012-10-15 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Neoplasms, Urinary Bladder
Keywords: Patients; Tumor antigens; Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cancer Group
  Interventions: Other: Data acquisition and analysis

INTERVENTIONS:
Other: Data acquisition and analysis — Tumor tissue samples submitted for analysis together with a form containing clinical data previously collected and archived from patients with bladder cancer.

SUMMARY:
This study aims to analyze the incidence of expression of MAGE-A3, MAGE-C2, NY-ESO-1, LAGE-1, WT1 and PRAME tumor antigens in cancer tissue from patients with pathologically demonstrated bladder cancer.

DETAILED DESCRIPTION:
There will be no procedure(s) or treatment(s) carried out on patients. All data and samples will be taken from those already stored at the investigation sites. Clinical data collected will include patient demographics (age, gender), Tumor, Node, Metastasis (staging system) [TNM stage], and histopathologic description only. Strict anonymity of patient data will be maintained.

This retrospective study is based upon the analysis of archived formalin-fixed paraffin-embedded tissue samples and patient-related data already available at the investigational site.

ELIGIBILITY:
Inclusion Criteria:

For inclusion of a tissue sample, all of the following criteria must be met:

* The patient had pathologically proven bladder cancer (any stage).
* All the data required are available from patient's records.

There are no restrictions regarding operative technique (cystectomy or cystoscopy).

- Many patients may no longer be alive, or no longer be in contact with the investigation sites. Thus, patients will not be required to give their informed consent before inclusion in the study.

Exclusion Criteria:

* Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously collected samples and data of patients with pathologically demonstrated bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2008-01-15 (Actual); Primary Completion 2008-01-15 (Actual); Study Completion 2008-01-15 (Actual)

PRIMARY OUTCOMES:
To determine the gene expression of MAGE-A3, MAGE-C2, NY-ESO-1, LAGE-1, WT1 and PRAME antigens in pathologically demonstrated bladder cancer. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leuven, Belgium

REFERENCES:
- [Derived] Lerut E, Van Poppel H, Joniau S, Gruselle O, Coche T, Therasse P. Rates of MAGE-A3 and PRAME expressing tumors in FFPE tissue specimens from bladder cancer patients: potential targets for antigen-specific cancer immunotherapeutics. Int J Clin Exp Pathol. 2015 Aug 1;8(8):9522-32. eCollection 2015. PMID 26464715